CLINICAL TRIAL: NCT01650675
Title: Indirect Assessment and Intervention for Perinatal Drug Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steven J. Ondersma, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: R01DA029050 (NIH); R01DA029050 (NIH)
Record Dates: First submitted 2012-07-13; First posted 2012-07-26 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Drug Abuse
Keywords: pregnancy; screening; motivation
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Participants randomized into the control condition complete assessment and a time-matched interactive session on infant nutrition.
  Interventions: Behavioral: Nutrition time control/placebo intervention
- Indirect intervention (Experimental): Participants in this condition review a short series of parenting strengths that benefit infants, and are invited to consider their current status in each area. This list includes factors associated with drug use (e.g., safety, emotional health) as well as substance use itself.
  Interventions: Behavioral: WIDUS computer-delivered, indirect brief intervention

INTERVENTIONS:
Behavioral: WIDUS computer-delivered, indirect brief intervention — A single 20-minute interactive computer-delivered intervention designed to promote motivation to change drug use and risky sexual behavior, if any, without presuming those risks to be specifically present.
  Arms: Indirect intervention
Behavioral: Nutrition time control/placebo intervention — This time-control intervention, designed in part to help promote RA blinding as to participant condition, focuses on proper infant nutrition using a computer-delivered, interactive format and videos.
  Arms: Control

SUMMARY:
The purpose of this study is to assess the validity of an indirect computer-delivered screener for drug use and assess the efficacy of a computer-delivered brief intervention with urban post-partum women at-risk for substance abuse and HIV during the post-partum period.

DETAILED DESCRIPTION:
Two factors limit the potential of brief interventions for the reduction of substance abuse and HIV risk. First, the ability to conduct such interventions is dependent upon willingness to disclose drug use and risky sexual behaviors. This is a significant obstacle given evidence that as few as half of drug-positive individuals-particularly women in the perinatal period-report that use. Second, there are logistic and financial obstacles to implementing even brief intervention programs, particularly with regard to time, training and provider willingness. In response to these limitations, and with NIDA support (DA018975), the Parent Health Lab at the Wayne State University School of Medicine developed and validated a sensitive indirect screener that evaluates correlates of illicit drug use rather than drug use itself. The Lab also developed a brief computer-delivered intervention designed to build change motivation without presuming the presence of risks to accompany the screener. This intervention demonstrated excellent feasibility and acceptability in Phase I testing. Following NIDA's Stage Model of Behavioral Therapy Development, the proposed study will take the next step of validating the computer-delivered indirect screening and intervention process in a Phase II/Stage IIb trial with women determined to be at risk by the indirect drug use screener. In addition, given that 47.8% of the prior sample's participants had an STI at some point in their lives, the proposed study will also further expand the existing focus on HIV risk. Specifically, we plan to: (a) continue development and validation of the WIDUS screener via concomitant collection of WIDUS protocols and hair/urine samples, as well as by building its ability to indirectly predict HIV risk; (b) revise and upgrade the draft indirect intervention based on expert and participant informant feedback; (c) recruit 500 at-risk women from an urban obstetric hospital; and (d) randomly assign participants into intervention and control conditions, with blinded follow-up assessments at 3- and 6-months. If proven efficacious, this logistically feasible, replicable, and low-cost approach could allow a dramatic increase in the reach--and therefore the population impact--of brief interventions for drug use among at-risk post-partum women. Further, any impact on maternal drug use would be further multiplied by indirect effects on the at-risk child.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* able to communicate in English
* recently gave birth to healthy infant

Exclusion Criteria:

* received narcotic pain medication in past 3 hours
* no sleep since giving birth
* infant deceased or in intensive care
* psychosis or other clear cognitive impairment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2012-06; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of drug using days | since last research visit; up to 90 days prior to current evaluation
  Drug use over past 90 days will be measured at a 3 and 6-month follow-up by self-report, hair, and urine analysis.
Change from Baseline HIV and other STI risk at 3 months | since last research visit; up to 90 days from baseline visit
  Self-report of risky sexual and/or injection drug use that could place participants at risk of HIV and other STIs
Change from Baseline in HIV and Other STI Risk at 6 months | since last research visit; up to 180 days since baseline visit
  Self-report of risky sexual and/or injection drug use that could place participants at risk of HIV and other STIs

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Ondersma, Ph.D., Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States